CLINICAL TRIAL: NCT00089947
Title: Randomized, Prospective, Phase 2 Study Comparing Thymoglobulin in a Rapid Discontinuation of Corticosteroids Protocol With Standard Corticosteroid Therapy in Living Donor Renal Transplantation Using Mycophenolate Mofetil and Tacrolimus Maintenance Therapy
Brief Title: A Study to Evaluate the Effect of Thymoglobulin and Reduced Doses of Steroids to Prevent Renal Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-101-1025
Record Dates: First submitted 2004-08-18; First posted 2004-08-20 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Renal Transplantation; Graft Rejection
Keywords: Anti-T cell antibodies; Living Donor Renal Transplantation; Acute Renal Allograft Rejection; Induction Therapy with Reduction of Calcineurin inhibitors
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum

INTERVENTIONS:
Drug: Thymoglobulin [Anti-Thymocyte Globulin (Rabbit)]

SUMMARY:
This study involves the use of a drug called Thymoglobulin, which is approved in the US to treat kidney transplant rejection and in Canada to treat and to prevent kidney transplant rejection.

This study will evaluate the effect of Thymoglobulin and reduced doses of steroids to prevent renal transplant rejection and will provide a basis for future evaluations of Thymoglobulin as an immunosuppressive agent to help prevent renal transplant rejection.

Subjects meeting all inclusion and exclusion criteria are eligible to participate in this study. In addition to standard treatment, study participants will receive either Thymoglobulin with rapid discontinuation of steroids or steroids per hospital standards for at least the first 90 days after transplant. The treatment assignment is random and is not chosen by the subject or their physician.

Subjects will be monitored during treatment with Thymoglobulin and during the transplant hospitalization. Additional subject monitoring occurs at Months 1, 3, 6 and 12 following the transplant.

Approximately 150 study subjects from 15-20 transplant centers in the United States will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult living donor renal transplant recipient
* Age greater than or equal to 18
* If female and of childbearing potential: a) must not be lactating; b) must have a negative serum B-human chorionic gonadotropin (HCG) test within 24 hours prior to Study Day 0 (Day of Transplant) and; c) must agree to practice an acceptable and reliable form of contraception during the study; and
* Signed informed consent

Exclusion Criteria:

* Human Leukocyte Antibody (HLA) identical matched living donor transplant recipient
* > 2 previous transplants
* Current panel reactive antibody (PRA) > 20%
* History of a positive cross-match with the donor
* Active donor or recipient serology positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis C virus (HCV)
* Loss of first kidney transplant in < 1 year
* History of noncompliance in clinical trial(s)
* History of chronic CS or immunosuppressive use except for inhaled CS to treat asthma
* Use of any investigational products during the 90 days prior to screening
* Requirement for multiple organ transplant
* Patient without a functioning urinary bladder prior to transplant (e.g. patients with self catheterization will be excluded)
* Known contraindication to administration of rabbit antithymocyte globulin
* Currently abusing drugs or alcohol
* In the opinion of the investigator, at high risk for poor compliance
* In the opinion of the investigator, has a significant medical or psychosocial problem or unstable disease state that warrants exclusion from the study. Examples of significant problems include, but are not limited to morbid obesity and severe cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
This study will evaluate the effect of Thymoglobulin and reduced doses of steroids to prevent renal transplant rejection, organ loss and death at 6 months.

SECONDARY OUTCOMES:
To evaluate patient kidney function after transplantation and the overall safety of Thymoglobulin in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (19):
- United States (19):
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Keck USC School of Medicine, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - University of California, San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Oschner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Texas Transplant Institute, San Antonio, Texas
  - Medical College of Virginia, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Thymoglobulin® — http://www.thymoglobulin.com/home/thymo_pdf_pi.pdf